CLINICAL TRIAL: NCT01226199
Title: The Expression of TLR2 and TLR4 in the Lung of COPD Patients
Brief Title: The Expression of TLR2 and TLR4 in the Lung of Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Sei Won Lee/ Assistant Professor, Seoul National University Bundang Hospital
Other Study IDs: TLR2 and TLR4 in COPD tissue
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Smoking; COPD
MeSH Terms: conditions — Smoking; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lung tissues are retained till the study ends.
Oversight: Data Monitoring Committee: No

SUMMARY:
Smoking is the most important risk factor of COPD, but only a fourth of smokers had COPD in their life. There are also healthy smokers without evidence of COPD. Investigators hypothesize that innate immunity may affect this difference between COPD patients and healthy smokers, because TLR4 is the receptor of LPS, which is the one of important substance in cigarette. Investigators will measure TLR2 and TLR4 expression in lung tissue of patients whose lung will be resected. Investigators will compare the level of expression between COPD patients and healthy smokers.

ELIGIBILITY:
Inclusion Criteria:

* All patients who will have lung resection for the therapeutic cause.

Exclusion Criteria:

* Patients who do not agree with our study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who will have lung resection for the therapeutic cause.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Gyeongi, South Korea